CLINICAL TRIAL: NCT05611073
Title: Maximizing Visual Outcomes With Eyhance IOLs
Status: Completed | Type: Observational
Sponsor: Berkeley Eye Center (Other)
Responsible Party: Sponsor
Other Study IDs: JMM-1261
Record Dates: First submitted 2022-07-12; First posted 2022-11-09 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pseudophakia
Keywords: Eyhance; Pseudophakia
MeSH Terms: conditions — Pseudophakia | interventions — Visual Acuity; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Distance with Minimal Intermediate Visual Acuity Group: Patients with bilateral implantation of Eyhance IOLs. And defined by BCDVA of 0.1 logMAR or better but a DCIVA of 0.4 logMAR or worse.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Biometric Data Collection; Other: Patient Questionnaire
- Distance with Enhanced Intermediate/Near Visual Acuity Group: Patients with bilateral implantation of Eyhance IOLS. And defined by BCDVA of 0.1 logMAR or better and a DCIVA of 0.3 logMAR or better.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Biometric Data Collection; Other: Patient Questionnaire

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Measurement of distance, intermediate and near visual acuity.
Diagnostic Test: Biometric Data Collection — Measurement of biometric data will be obtained from the Zeiss IOL Master 700, Atlas 9000, and the iTrace.
Other: Patient Questionnaire — Patients will complete a Patient Questionnaire to determine their level of spectacle independence and visual acuity satisfaction.

SUMMARY:
This is a non-interventional prospective, single center, bilateral, non-randomized, open-label, observational clinical study. All patients will have had bilateral implantation of an Eyhance IOL at the time of cataract surgery. These patients will then be compared to assess which patient biometric properties (such as spherical aberration, q value, pupil size, etc.) lead to an overall increase in near or intermediate vision as well as overall patient satisfaction.

DETAILED DESCRIPTION:
This is a non-interventional prospective, single center, bilateral, non-randomized, open-label, observational clinical study. All patients will have had bilateral implantation of an Eyhance IOL at the time of cataract surgery. These patients will then be assessed in the 1-6-month post-operative period. Patients will be grouped into two arms: "distance with minimal intermediate" and "distance with enhanced intermediate/near" based on mean photopic binocular BCDVA and DCIVA (at 66 cm) of patients with bilateral Eyhance IOLs corrected to plano sphere. The "distance with minimal intermediate" group is defined by BCDVA of 0.1 logMAR or better but a DCIVA of 0.4 logMAR or worse. The "distance with enhanced intermediate/near" is defined by BCDVA of 0.1 logMAR or better and a DCIVA of 0.3 logMAR or better. In addition to binocular BCDVA and DCIVA, monocular measurements will be obtained as well. The two groups will be compared to assess which patient biometric properties (such as spherical aberration, q value, pupil size, etc.) lead to an overall increase in near or intermediate vision as well as overall patient satisfaction. Biometric data will be obtained from the Zeiss IOL Master 700, Atlas 9000, and the iTrace.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 40 years of age having already undergone uncomplicated cataract removal by phacoemulsification with a clear corneal incision in both eyes.
2. Implantation of bilateral Eyhance IOLs (DIB00/DIU***).
3. Able to comprehend and willing to sign informed consent and complete all required testing procedures.
4. Best Corrected Distance Visual Acuity (BCDVA) projected to be 0.10 logMAR (Minimum Angle of Resolution) or better.
5. Clear intraocular media.
6. Minimum of two weeks post YAG capsulotomy to treat PCO

Exclusion Criteria:

1. Any corneal abnormality, other than regular corneal astigmatism (as determined by pre-operative testing) that in the opinion of the investigator would confound the outcome(s) of the study.
2. Any complication during cataract surgery (capsular tear, vitrectomy, etc.).
3. History of or current retinal conditions or predisposition to retinal conditions.
4. Amblyopia or strabismus in either eye.
5. History of or current anterior or posterior segment inflammation of any etiology.
6. Any form of neovascularization on or within the eye.
7. Glaucoma (uncontrolled or controlled with medication).
8. Optic nerve atrophy.
9. Subjects with diagnosed degenerative eye disorders.
10. Postoperative CDVA worse than 0.10 logMAR (20/25 snellen).
11. Subjects who have an acute or chronic disease or illness that would confound the results of this investigation in the opinion of the investigator (e.g. immunocompromised, connective tissue disease, clinically significant atopic disease, etc.).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with healthy eyes and uncomplicated bilateral implantation of Eyhance IOLs.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Started | 49 | 61
Completed | 49 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group | Total
Number analyzed (Participants) | 49 | 61 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (6.5) | 69.8 (7.3) | 69.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 24 | 58
  Male | 15 | 37 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Two Groups Categorized by "Distance With Minimal Intermediate" and "Distance With Enhanced Intermediate/Near" Based on Mean Photopic Binocular BCDVA of Patients With Bilateral Eyhance IOLs Corrected to Plano Sphere.
Description: To compare two groups categorized by "distance with minimal intermediate" and "distance with enhanced intermediate/near" based on mean photopic binocular BCDVA of patients with bilateral Eyhance IOLs targeted corrected at plano sphere.
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
logMAR | 0.03 (0.04) | 0.01 (0.02)

2. Primary Outcome: Comparison of Two Groups Categorized by "Distance With Minimal Intermediate" and "Distance With Enhanced Intermediate/Near" Based on Mean Photopic Binocular DCIVA (at 66 cm) of Patients With Bilateral Eyhance IOLs Corrected to Plano Sphere.
Description: To compare two groups categorized by "distance with minimal intermediate" and "distance with enhanced intermediate/near" based on mean photopic binocular DCIVA (66 cm) of patients with bilateral Eyhance IOLs targeted corrected at plano sphere.
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
logMAR | 0.30 (0.07) | 0.12 (0.07)

3. Secondary Outcome: Determine if Any Statistically Significant Differences in Pupil Size Exists Between the Two Groups.
Description: To determine if any statistically significant differences in pupil size exists between the two groups that may allow for pre-operative recognition of those patients who could have enhanced benefits of the Eyhance IOL. This will require multiple regression analysis given the large number of variables.
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
Number analyzed (eyes) | 98 | 122
mm | 4.16 (0.77) | 3.64 (0.77)

4. Secondary Outcome: Spherical Aberration Between Groups
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: microns (µm)
Units Other Than Participants: eyes
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
Number analyzed (eyes) | 98 | 122
microns (µm) | 0.29 (0.16) | 0.31 (0.15)

5. Secondary Outcome: Q Value Between Groups.
Description: Q-value is an assessment of corneal asphericity.
  * A value of 0 indicates a cornea that is perfectly spherical
  * A value between -1 and 0 indicates a cornea that is shaped more like a football
  * A value between 0 and 1 indicates a cornea that is shaped more like a dish
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: Q value
Units Other Than Participants: eyes
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
Number analyzed (eyes) | 98 | 122
Q value | -0.34 (0.23) | -0.31 (0.18)

6. Secondary Outcome: Biometric Data (Anterior Chamber Depth and Axial Length) Between Groups.
Description: To determine if any statistically significant differences in biometric data exists between the two groups that may allow for pre-operative recognition of those patients who could have enhanced benefits of the Eyhance IOL. This will require multiple regression analysis given the large number of variables.
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
Number analyzed (eyes) | 98 | 122
mm
  Anterior Chamber Depth | 3.25 (0.32) | 3.19 (0.41)
  Axial Length | 24.33 (1.36) | 24.34 (1.52)

7. Other Pre Specified Outcome: Comparison of a Patient Satisfaction Survey Between the Two Groups to Assess for Subjective Differences in Everyday Life. Patient's Answers Will be on a Scale Between Always and Never, Where Never Shows a Better Patient Outcome.
Description: Comparison of a patient satisfaction survey between the two groups to assess for subjective differences in everyday life to determine if the enhanced vision plays a statistically significant difference in patient's perceived quality of vision or quality of life. Patient's answers will be on a scale between always and never, where never shows a better patient outcome.
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Measure: Number; unit: percentage of participants
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
Number analyzed (Participants) | 49 | 61
percentage of participants
  Never experiencing glare, halos, or starbursts. | 45 | 66
  Never using glasses for distance vision | 69 | 84
  Never using glasses for intermediate vision | 55 | 59
  Never using glasses for near vision | 24 | 30

ADVERSE EVENTS:
Time Frame: 1 day (between a minimum of 3 weeks postoperative up to 26 weeks post-operative)
Arm/Group | Distance With Minimal Intermediate Visual Acuity Group | Distance With Enhanced Intermediate/Near Visual Acuity Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/61
Other Adverse Events (participants affected / at risk) | 0/49 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT05611073/Prot_SAP_000.pdf